CLINICAL TRIAL: NCT04913480
Title: A Multi-centre Single-arm Phase II Study on Durvalumab (MEDI 4736) With Stereotactic Body Radiation Therapy (SBRT) in Patients With Inoperable/Unresectable Hepatocellular Carcinoma
Brief Title: SBRT and Durvalumab for Inoperable/Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Victor H.F. Lee, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 19-655
Record Dates: First submitted 2021-05-22; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Immune checkpoint inhibitor; Stereotactic body radiation therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Combination of stereotactic body radiation therapy and immune checkpoint inhibitor for inoperable/unresectable hepatocellular carcinoma
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab and stereotactic body radiation therapy (Experimental): 1. Durvalumab 750mg intravenous infusion once every 2 weeks for 26 cycles, starting 1 week before commencement of stereotactic body radiation therapy
  2. Stereotactic body radiation therapy of 27.5Gy to 50Gy in 5 fractions to the liver tumors delivered over 5 to 14 days
  Interventions: Drug: Durvalumab; Radiation: Stereotactic body radiation therapy

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 750mg intravenous infusion once every 2 weeks for 26 cycles
  Other Names: MEDI4736
Radiation: Stereotactic body radiation therapy — Stereotactic body radiation therapy of 27.5Gy to 50Gy in 5 fractions to the liver tumors delivered over 5 to 14 days.
  Other Names: Stereotactic body radiotherapy

SUMMARY:
The investigators propose a phase II single-arm study on using stereotactic body radiation therapy in combination with durvalumab for inoperable/unresectable hepatocellular carcinoma. In addition, the investigators will also measure the change in number and intensity of PD-L1-positive circulating tumor cells before and after stereotactic body radiation therapy and durvalumab and evaluate their correlation with treatment response.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the commonest solid malignancies in Asia Pacific region, primarily because of high incidence of hepatitis B infection in this locality. Resection or liver transplantation is the standard treatment for operable/resectable disease. However more than 50% of HCC are inoperable, primarily because of poor liver function, limited normal liver reserve and advanced disease beyond resectability. Locoregional treatment including transarterial chemoembolization (TACE), percutaneous ethanol injection (PEI), radiofrequency ablation (RFA) and recently radio-embolization are acceptable options. However the response rate was just between 30-80% treated with these modalities. Also some patients are contraindicated to these local therapies. For instance, those who have poor liver function (Child-Pugh B) or have their tumors showing portal vein invasion/thrombosis are contraindicated to TACE. Those who had their tumors close to adjacent critical organs e.g. liver, stomach, duodenum, small bowel and gallbladder, etc were not candidates for RFA or percutaneous ethanol injection. In addition, those who had tumors >4cm or close to major vessels have high local recurrence after RFA. Stereotactic body radiation therapy (SBRT), with the use of highly conformal and precision radiation techniques with real-time tracing of patient and tumor position so as to offer a high radiation dose to the tumors while sparing the adjacent critical organs from necessary radiation.

Previous preclinical studies suggested synergism of anti-tumor activity between radiation therapy and immune checkpoint inhibitors. Immune checkpoint inhibitors are now comprehensively and extensively tested in combination with radiotherapy (RT) as well (NCT01935921, NCT01860430). It has been recently known that RT increases the expression of the major histocompatibility complex (MHC). In turn, the MHC class-I restricted tumor antigen-specific cells elicited by RT will upregulate interferons in the tumors. This radiation-induced local inflammation and tumor-specific effector T cells will provide an additional mechanism for tumor control by modification of the tumor vasculature. In addition, RT will increase dendritic cell surface antigen presentation to T cells and production of cytokines leading to recruitment and activation of leucocytes from peripheral blood and extravasation to tumor parenchyma. These are part of the mechanisms of abscopal effect, a phenomenon where the tumors at the sites far away from the irradiated sites also regress after localized radiotherapy. Having learnt from the pivotal PACIFIC trial on the use of consolidation therapy with durvalumab (anti-PD-L1 monoclonal antibody) which confirmed the efficacy and safety of combination of chemoradiation and immunotherapy for stage III non-small-cell lung cancer, it is prime time to consider incorporation of immune checkpoint inhibitors into concurrent chemoradiation for other solid tumors like HCC.

In view of the promising activity of SBRT and immune checkpoint inhibitors for HCC, we propose a phase II single-arm study on using durvalumab in combination with SBRT for inoperable/unresectable HCC. Recruited patients with receive durvalumab 750mg intravenously every 2 weeks, starting 1 week before SBRT, for a total of 26 cycles (1 year).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or radiologically confirmed HCC. For radiological diagnosis of HCC, a contrast-enhanced computed tomography or magnetic resonance imaging is mandatory to demonstrate the early arterial enhancement in arterial phase and contrast washout in the porto-venous phase on the imaging.
2. Inoperable or unresectable non-metastatic HCC (in the form of tumor resection or liver transplantation) amenable to stereotactic body radiation therapy given in 5 fractions. Prior locoregional therapy including radiofrequency ablation, transarterial chemoembolisation, radioembolisation is allowed provided that radiologically progressive disease is demonstrated following these locoregional therapies.
3. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorisation (e.g. Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
4. Be >/= 18 years of age on day of signing informed consent.
5. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
6. A stage C or earlier HCC based on Barcelona Clinic Liver Cancer (BCLC) staging system.
7. A Child-Pugh of 7 or less.
8. Demonstrate adequate organ function as defined in Inclusion Criteria 7, all screening labs should be performed 28 days prior to study registration up to the first dose of study drug.
9. Adequate serum hematological functions defined as:

   * Absolute neutrophil count (ANC) ≥1.0 x 10^9/l
   * Platelet ≥50 x 10^9/l
   * Hemoglobin ≥9 g/dL

   Adequate serum biochemistry functions defined as:
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). <<This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.>>
   * Serum aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤2.5 times of institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5 times of ULN
   * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
10. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 times of ULN unless subject is receiving anticoagulant therapy as long as PT or activated partitional thromboplastin time (APTT) is within therapeutic range of intended use of anticoagulants. APTT ≤1.5 times of ULN unless subject is receiving anticoagulant therapy as long as PT or APTT is within therapeutic range of intended use of anticoagulants.
11. Female subject of childbearing potential should have a negative urine or serum pregnancy within 24 hours of study enrollment up to administration of the dose of study drug. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 31 weeks after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
13. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 31 weeks after the last dose of study therapy.
14. We will allow prior radiation to other sites, with no washout period, prior to study entry as long as the high dose regions of the prior and proposed radiation fields do not overlap. In patients where the prior high dose area would overlap with the high dose area of the intended radiation, a 4 month washout period will be required. The safety of such treatment will be at discretion of the treating radiation oncologist.
15. Prior central nervous system (CNS) radiation is allowed as long as cumulative radiation doses do not exceed tolerance of critical structures as judged by the treating radiation oncologist.
16. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
17. Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment or 5 half-lives, whichever is shorter.
2. Has a diagnosis of severe active scleroderma, lupus, other rheumatologic or autoimmune disease within the past 3 months before study recruitment. Patients with a documented history of clinically severe autoimmune disease or a syndrome requiring systemic steroids or immunosuppressive agents will not be allowed on this study. Subjects with vitiligo or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections are not excluded from the study. Subjects with hypothyroidism stable on hormone replacement are not excluded from this study.
3. Has had a prior monoclonal antibody, immunotherapy or immune checkpoint inhibitors before recruitment into this study .
4. Has had prior chemotherapy or targeted small molecule therapy (including sorafenib or other anti-vascular endothelial growth factor inhibitor) within 3 weeks prior to administration of the study drug or who has not recovered (i.e., ≤Grade 1 or at baseline) from adverse events due to a previously administered agent. *Note: Subjects with permanent ≤ Grade 2 toxicities (e.g. neuropathy) or toxicities corrected through routine medical management (e.g. thyroid replacement for hypothyroidism), are an exception to this criterion and may qualify for the study. *Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. *Note: Subjects with ≤ Grade 2 amylase or lipase elevations abnormalities that have no corresponding clinical manifestations (e.g. manifestation of pancreatitis), are an exception to this criterion and may qualify for the study.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, indolent lymphomas, or in situ cervical cancer that has undergone potentially curative therapy
6. Has a history of prior solid organ transplants with or without any episodes of graft-versus-host disease.
7. Has a history of allogeneic bone marrow transplantation and peripheral stem cell rescue, with or without any episodes of graft-versus-host disease.
8. Has clinically significant or symptomatic ascites requiring either diuretic therapy or paracentesis.
9. Has known active extra-hepatic metastases. Patients with treated extra-hepatic metastases which are stable and not requiring any systemic treatment for ≥ 4 weeks are eligible.
10. Has known carcinomatous meningitis (also known as leptomeningeal carcinomatosis).
11. Has an active infection requiring intravenous systemic therapy or hospital admission.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality, including psychiatric or substance abuse disorder, that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 31 weeks after the last dose of trial treatment.
14. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). Routine checking for Anti-HIV1 or Anti-HIV2 is not mandatory.
15. Untreated hepatitis B infection. Patients with chronic hepatitis B infection (defined as HBsAg positive) are eligible if they have started anti-viral therapy for at least 1 month and is continuing anti-viral treatment throughout the whole duration of this study.
16. Has received a live vaccine 30 days prior to the first dose of trial treatment.
17. Has experienced Grade 4 toxicity on treatment with prior radiation.
18. Has experienced Grade 3-4 intracranial toxicity (hypophysitis or CNS toxicity) with either prior intracranial radiation, anti programmed cell death-1 (PD-1), or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitor therapy.
19. Is taking >4mg/day of dexamethasone or its equivalent at the start of immunotherapy or has required >4mg/day of dexamethasone or its equivalent for 3 consecutive days within 1 week of starting treatment.
20. Allergies and adverse drug reaction to the following: History of allergy to study drug components; History of severe hypersensitivity reaction to any monoclonal antibody.
21. Prior systemic therapy utilizing an anti CTLA-4 or PD-1/PD-L1 agent or other forms of immunotherapy.
22. Has had prior radiation therapy (defined as >1Gy) to the area planning to be treated with SBRT.
23. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
24. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
25. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

(A) Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) (B) Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent (C) Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 1 year | 12 months
  Progression-free survival at 1 year

SECONDARY OUTCOMES:
Best objective response | 36 months
  Best objective response
Local control rate | 36 months
  Local control rate
Liver failure-free rate | 36 months
  Liver failure-free rate
Overall survival | 36 months
  Overall survival
Incidence of treatment-related side effects | 36 months
  Incidence of treatment-related side effects as determined by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Changes in PD-L1 and PD-1 positive circulating tumor cells before and after stereotactic body radiation therapy and durvalumab | 36 months
  Changes in PD-L1 and PD-1 positive circulating tumor cells before and after stereotactic body radiation therapy and durvalumab

CONTACTS AND LOCATIONS:
Overall Officials: Victor Ho Fun Lee, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.